CLINICAL TRIAL: NCT00290836
Title: An Open, Randomised, Prospective, Single-centre Phase IV Trial to Assess Efficacy and Safety of TachoComb H Versus Standard Surgical Treatment (i.e. Suture) in Patients Undergoing Prostatectomy
Brief Title: Assess Efficacy and Safety of TachoComb H vs. Standard Surgical Treatment (i.e. Suturing) in Patients Undergoing Prostatectomy (TC-017-AU)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-017-AU
Record Dates: First submitted 2005-12-16; First posted 2006-02-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Control of Local Bleeding in Patients Undergoing Prostatectomy.
MeSH Terms: interventions — Fibrinogen; Thrombin; Aprotinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Human fibrinogen/thrombin and bovine aprotinin (TachoComb H)

SUMMARY:
The overall objective is to compare efficacy and safety of TachoComb H versus standard surgical treatment for the control of local bleeding in patients undergoing prostatectomy. Specific objectives include the comparison between test treatments for intraoperative haemostatic efficacy as well as for post-operative blood loss to be assessed by haemoglobin and haematocrit concentration of drainage fluid.

ELIGIBILITY:
Inclusion Criteria:

1. has the subject given informed consent according to local requirements before any trial related activies? A trial related activity is any procedure that would not have been performed during the routine management of the subject.
2. Is the subject 18 years of age or above ?
3. Is the subject planned for a radical prostatectomy for prostate cancer (cT3)?

   After prostate resection and primary haemostatic treatment
4. is only minor (i.e. oozing) or moderate haemorrhage persisting after primary surgical haemostatic procedures of the major vessels (no pulsating arterial haemorrhage and/or major venous bleeding)?

Exclusion:

At pre-operative screen

1. Is there anamnestic or laboratory evidence of coagulation disorders including haemophilia A or B and von Willebrand disease ?
2. Has the patient a history of allergic reactions after application of human fibrinogen, human thrombin, bovine aprotinin and/or collagen of any origin?
3. Is the patient undergoing an emergency operation?
4. Did the patient participate in a clinical trial less than 30 days prior to inclusion in present trial?
5. Does the patient participate in a clinical trial concomitantly with present trial?

   After tumour resection and primary haemostatic treatment
6. Has any serious surgical complication occurred?
7. Has any fibrin glue haemostatic (including any type of TachoComb) been used before randomisation?

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy: Is the percentage of patients/treatment group in which efficient intra-operative haemostasis is achieved within 10 minutes after applying test treatment according to randomisation after primary surgical haemostasis.

SECONDARY OUTCOMES:
Efficacy:
Haemoglobin concentration of drainage fluid on day 1 after surgery.
Haemotocrit concentration of drainage fluid on day 1 after surgery.
Volume of drainage fluid on day 1 after surgery.
Incidence of post-operative haematoma at removal site at day 2 after surgery (sonography).
Incidence of tumour positive resection margin proven by histology (discharge).
Reporting of occurrence of urinary incontinence (discharge, 3 months +/- 10 days (and optional 12 months +/- 30 days) after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark